CLINICAL TRIAL: NCT04813432
Title: Low Dose Multi-arterial Phase CT Imaging for Improved Detection of Liver Tumors and Pancreatic Masses
Brief Title: Multiple Arterial Phase Computed Tomography Examination to Improve Detection of Tumors in the Liver and Pancreas
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Katharina Brehmer, principal investigator, Karolinska Institutet
Other Study IDs: EPN Diarienr. 2018/859-31
Record Dates: First submitted 2020-11-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Contrast Media; Computed Tomography; Imaging; Pancreatic Cancer; Hepatic Cancer
Keywords: computed tomography; CT angiography; hepatic imaging; pancreatic imaging; hepatocellular cancer; pancreatic adenocarcinoma; liver; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Computed Tomography of the Abdomen — Multi-phasic CT scan of the abdomen: 1 low dose unenhanced scan + 10 low dose arterial perfusion scans + 1 portal-venous phase scan + 1 delayed phase scan.
  Bolus-tracking threshold in abdominal aorta = 160 HU. Delay of first arterial scan 5 sec after bolus-tracking threshold has been reached; and then 1 scan every 3 sec until 35 sec after threshold.
  Contrast media (CM) protocol: fixed injection duration: 25 sec, body weight-adjusted CM volume: 750 mgI/kg bodyweight (max 80 kg women, 100kg men), Iomeron 400mgI/ml.
  Image-reconstruction: Motion-correction, noise-reduction and fusion of the best arterial time points to reconstruct one optimally timed early and one optimally timed late arterial phase.

SUMMARY:
To examine inter-subject variations of optimal late arterial phase contrast-enhancement defined as the greatest difference in contrast attenuation of hepatocellular carcinoma (HCC) compared to background liver parenchyma resp. pancreatic lesions compared to pancreatic parenchyma. To evaluate which time-points best depict an optimal late arterial phase.

DETAILED DESCRIPTION:
Background: Many previous studies have analyzed and proposed different strategies to achieve optimal contrast timing and enhancement in the late arterial phase to best depict arterialized lesions in the liver and hypoattenuating tumors in the pancreas(1-12). But even with the use of state-of-the-art protocols, inter-subject variations of optimal contrast enhancement in liver lesions and pancreas parenchyma are still very common. The aim of this study is to first analyze these alterations and to, secondly, use the newly gained knowledge to design a dose-neutral multiple arterial phase protocol. An optimized arterial phase protocol might improve the detection of hepatocellular carcinoma (HCC) and/or pancreatic adenocarcinoma.

Purpose: To measure when the greatest difference in attenuation occurs in HCC compared to background liver parenchyma resp. in pancreatic lesions vs. pancreatic parenchyma. To describe the inter-subject variation of these enhancement times and to evaluate at which time-points an optimal late arterial phase can be achieved. The investigators will use the perfusion scanning technique, bolus-tracking and high body-weight-adjusted volumes of contrast media (CM).

Anticipated results: The aim is to find the best time points for optimal CM-enhancement in HCC lesions and pancreas parenchyma. The results will show the extent of the inter-subject temporal enhancement differences and will be used to design an optimized late arterial phase protocol for clinical practice and future studies.

ELIGIBILITY:
Inclusion Criteria:

* patients, who are scheduled for a multiphasic liver or pancreas CT because of known or suspected malignancy in the liver or pancreas.

Exclusion Criteria:

* below 50 years of age, contrast media allergy or decreased kidney function

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 consecutive patients, who are scheduled for a multiphasic liver or pancreas CT because of known treatment naïve or suspected HCC or pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Peak enhancement values measured in Hounsfield units(HU) in abdominal aorta. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in abdominal aorta.
Peak enhancement times measured in seconds in abdominal aorta. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in abdominal aorta.
Peak enhancement values measured in Hounsfield units(HU) in celiac trunc. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in celiac trunc.
Peak enhancement times measured in seconds in celiac trunc. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in celiac trunc.
Peak enhancement values measured in Hounsfield units(HU) in superior mesenteric artery (SMA). | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in SMA.
Peak enhancement times measured in seconds in superior mesenteric artery (SMA). | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in SMA.
Peak enhancement values measured in Hounsfield units(HU) in hepatic artery. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in hepatic artery.
Peak enhancement times measured in seconds in hepatic artery. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in hepatic artery.
Peak enhancement values measured in Hounsfield units(HU) in portal vein. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in portal vein.
Peak enhancement times measured in seconds in portal vein. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in portal vein.
Peak enhancement values measured in Hounsfield units(HU) in pancreas parenchyma. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in pancreas parenchyma.
Peak enhancement values measured in Hounsfield units(HU) in pancreatic lesions. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in pancreatic lesions.
Peak enhancement times measured in seconds in pancreas parenchyma. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in pancreas parenchyma.
Peak enhancement times measured in seconds in pancreatic lesions. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in pancreatic lesions.
Peak enhancement values measured in Hounsfield units(HU) in liver parenchyma. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in liver parenchyma.
Peak enhancement values measured in Hounsfield units(HU) in hepatic lesions. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in hepatic lesions.
Peak enhancement times measured in seconds in liver parenchyma. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in liver parenchyma.
Peak enhancement times measured in seconds in hepatic lesions. | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  Creation of time attenuation curves (TAC) in hepatic lesions.
highest enhancement difference between a hepatic lesion and background liver parenchyma | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  To measure the highest enhancement difference in Hounsfield units(HU) between a hepatic lesion and background liver parenchyma
time-point of highest enhancement difference between a hepatic lesion and background liver parenchyma | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  To depict the time-point of the highest enhancement difference between a hepatic lesion and background liver parenchyma by comparing their tissue attenuation curves
highest enhancement difference between a pancreatic lesion and background pancreatic parenchyma | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  To measure the highest enhancement difference in Hounsfield units(HU) between a pancreatic lesion and background pancreas parenchyma
time-point of highest enhancement difference between a pancreatic lesion and background pancreatic parenchyma | at the time of intervention (= Multi-phasic CT scan of the abdomen)
  To depict the time-point of the highest enhancement difference between a pancreatic lesion and background pancreas parenchyma by comparing their tissue attenuation curves

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Brehmer, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Radiology Department, Karolinska Huddinge university hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bae KT. Intravenous contrast medium administration and scan timing at CT: considerations and approaches. Radiology. 2010 Jul;256(1):32-61. doi: 10.1148/radiol.10090908. PMID 20574084
- [Background] Kondo H, Kanematsu M, Goshima S, Miyoshi T, Shiratori Y, Onozuka M, Moriyama N, Bae KT. MDCT of the pancreas: optimizing scanning delay with a bolus-tracking technique for pancreatic, peripancreatic vascular, and hepatic contrast enhancement. AJR Am J Roentgenol. 2007 Mar;188(3):751-6. doi: 10.2214/AJR.06.0372. PMID 17312064
- [Background] Bae KT, Heiken JP. Scan and contrast administration principles of MDCT. Eur Radiol. 2005 Dec;15 Suppl 5:E46-59. doi: 10.1007/s10406-005-0165-y. PMID 18637230
- [Background] Rengo M, Bellini D, De Cecco CN, Osimani M, Vecchietti F, Caruso D, Maceroni MM, Lucchesi P, Iafrate F, Paolantonio P, Ferrari R, Laghi A. The optimal contrast media policy in CT of the liver. Part I: Technical notes. Acta Radiol. 2011 Jun 1;52(5):467-72. doi: 10.1258/ar.2011.100499. Epub 2011 Mar 17. PMID 21498281
- [Background] Rengo M, Bellini D, De Cecco CN, Osimani M, Vecchietti F, Caruso D, Maceroni MM, Lucchesi P, Iafrate F, Palombo E, Paolantonio P, Ferrari R, Laghi A. The optimal contrast media policy in CT of the liver. Part II: Clinical protocols. Acta Radiol. 2011 Jun 1;52(5):473-80. doi: 10.1258/ar.2011.100500. Epub 2011 Mar 28. PMID 21498280
- [Background] Fleischmann D, Kamaya A. Optimal vascular and parenchymal contrast enhancement: the current state of the art. Radiol Clin North Am. 2009 Jan;47(1):13-26. doi: 10.1016/j.rcl.2008.10.009. PMID 19195531
- [Background] Delrue L, Blanckaert P, Mertens D, De Waele J, Ceelen W, Achten E, Duyck P. Variability of CT contrast enhancement in the pancreas: a cause for concern? Pancreatology. 2011;11(6):588-94. doi: 10.1159/000334547. Epub 2012 Jan 11. PMID 22237307
- [Background] Goshima S, Kanematsu M, Kondo H, Yokoyama R, Miyoshi T, Nishibori H, Kato H, Hoshi H, Onozuka M, Moriyama N. MDCT of the liver and hypervascular hepatocellular carcinomas: optimizing scan delays for bolus-tracking techniques of hepatic arterial and portal venous phases. AJR Am J Roentgenol. 2006 Jul;187(1):W25-32. doi: 10.2214/AJR.04.1878. PMID 16794136
- [Background] Heiken JP, Brink JA, McClennan BL, Sagel SS, Crowe TM, Gaines MV. Dynamic incremental CT: effect of volume and concentration of contrast material and patient weight on hepatic enhancement. Radiology. 1995 May;195(2):353-7. doi: 10.1148/radiology.195.2.7724752.
- [Background] Ichikawa T, Erturk SM, Araki T. Multiphasic contrast-enhanced multidetector-row CT of liver: contrast-enhancement theory and practical scan protocol with a combination of fixed injection duration and patients' body-weight-tailored dose of contrast material. Eur J Radiol. 2006 May;58(2):165-76. doi: 10.1016/j.ejrad.2005.11.037. Epub 2006 Jan 18. PMID 16417983
- [Background] Schueller G, Schima W, Schueller-Weidekamm C, Weber M, Stift A, Gnant M, Prokesch R. Multidetector CT of pancreas: effects of contrast material flow rate and individualized scan delay on enhancement of pancreas and tumor contrast. Radiology. 2006 Nov;241(2):441-8. doi: 10.1148/radiol.2412051107. Epub 2006 Sep 18. PMID 16982815
- [Background] Tang A, Billiard JS, Chagnon DO, Rizk F, Olivie D, Turcotte S, Chagnon M, Lepanto L. Optimal Pancreatic Phase Delay with 64-Detector CT Scanner and Bolus-tracking Technique. Acad Radiol. 2014 Aug;21(8):977-85. doi: 10.1016/j.acra.2014.04.004. PMID 25018069